CLINICAL TRIAL: NCT03706677
Title: FIRE AND ICE II Trial Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Collaborators: genae associates (CRO), Antwerp, Belgium (Unknown); King's College London (Other); Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MDT17037
Record Dates: First submitted 2018-09-17; First posted 2018-10-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Persistent Atrial Fibrillation; Atrial Arrhythmia
Keywords: Ablation; Cryoballoon; Radiofrequency
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Randomization 1:1 between Cryoballoon ablation and Radiofrequency ablation
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Single-blinded; participants will be blinded to the treatment group. Investigators will be blinded on study specific diagnostics used in the trial; Endpoint Review Committee will be blinded to the treatment group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRYO group (Active Comparator): Within the CRYO arm the ablation will be performed using the Arctic Front Advance Cardiac CryoAblation Catheter, including next generation systems as applicable and approved by Medtronic for the trial.
  Intervention performed: Cryoballoon ablation; Cryoballoon (Arctic Front Advance Cryoballoon)
  Interventions: Device: Cryoballoon (Arctic Front Advance Cryoballoon)
- RF group (Active Comparator): Within the RF arm the ablation will be performed using a catheter out of the ThermoCool Smarttouch catheter family, including next generation contact force systems as applicable.
  Intervention performed: Radiofrequency ablation; Radiofrequency Catheter (ThermoCool Smarttouch)
  Interventions: Device: Radiofrequency Catheter (ThermoCool Smarttouch)

INTERVENTIONS:
Device: Cryoballoon (Arctic Front Advance Cryoballoon) — Ablation using a Cryoballoon catheter (Arctic Front Advance Cryoballoon Cardiac Ablation Catheter)
  Arms: CRYO group
Device: Radiofrequency Catheter (ThermoCool Smarttouch) — Ablation using a Radiofrequency ablation catheter (ThermoCool Smarttouch catheter)
  Arms: RF group

SUMMARY:
The FIRE AND ICE II Trial (Pilot) is the pilot phase of a prospective, randomized, single-blinded, multi-center, interventional post-market clinical trial, comparing efficacy and safety of isolation of the pulmonary veins (PVI) using a Cryoballoon catheter or radiofrequency ablation with a ThermoCool® Smarttouch® catheter in subjects with persistent atrial fibrillation (AF).

DETAILED DESCRIPTION:
60 patients with persistent AF will be randomized 1:1 between Cryoballoon ablation and Radiofrequency ablation in the FIRE AND ICE II Trial Pilot at 5 clinical sites in Europe.

The data collected within the pilot phase will be reviewed and a decision on extending the trial with an extended number of patients and sites as main phase will be taken.

ELIGIBILITY:
Key Inclusion Criteria

* Documentation of symptomatic persistent AF (following the European Society of Cardiology (ESC) guideline 2016) defined as: Persistent AF - AF that lasts longer than 7 days, including episodes that are terminated by cardioversion, either with drugs or by direct current cardioversion, after 7 days or more
* Date of first diagnosis of persistent AF within the last 12 months preceding the date of screening
* Documented treatment failure or intolerance of at least one Class I or Class III antiarrhythmic drug

Key Exclusion Criteria

* Known pre-existing hemi-diaphragmatic paralysis
* Prior left atrial ablation or surgical procedure (including left atrial appendage closures)
* History of right atrial flutter, not ablated prior to enrollment
* Any cardiac surgery, myocardial infarction, percutaneous coronary intervention or coronary artery stenting which occurred within the 3 months before the eligibility assessment
* Unstable angina pectoris
* Primary pulmonary hypertension
* Any condition contraindicating chronic anticoagulation
* Any cerebral ischemic event (stroke or transient ischemic attack [TIA]) which occurred within the 6 months before the consent date
* Presence of any cardiac prosthetic valves
* Long-standing persistent AF lasting for ≥ 1 year (even when it is decided to adopt a rhythm control strategy)
* New York Health Association (NYHA) class III or IV heart failure and/or documented left ventricular ejection fraction (LVEF) < 40% measured by acceptable cardiac testing (e.g. TTE)
* Acute cardiac condition, including endocarditis, pericarditis or pericardial effusion
* Presence or likely implant of a permanent pacemaker, biventricular pacemaker or any type of implantable cardiac defibrillator (with or without biventricular pacing function) within 12 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Objective (not powered within pilot) (time to clinical treatment failure) | 12 Month
  To demonstrate that Cryo ablation is non-inferior to radiofrequency (RF) ablation with respect to time to clinical treatment failure, defined as recurrence of atrial arrhythmias or intervention for AF (a blanking period of three months will be maintained after the index procedure). The first documented recurrence of an episode of atrial arrhythmia after the blanking period lasting at least 30 seconds will be counted for the primary efficacy objective, as well as any intervention for AF with initiation after the blanking period.
Safety Objective (freedom from device and procedure related serious adverse events (SAEs)) | 12 Month
  To demonstrate that Cryo ablation is non-inferior to RF ablation with respect to freedom from device and procedure related serious adverse events (SAEs). The first device or procedure related serious adverse event with onset after start of the index ablation therapy will be used for the safety objective analysis.

SECONDARY OUTCOMES:
Assess acute procedural success (PVI) | 3 Month
  Acute procedural success is defined as successful electrical isolation of the pulmonary veins after the ablation procedure as assessed via a diagnostic catheter.
Assess quality of life: EQ-5D-5L | 12 Month and 36 Month
  The EQ-5D-5L and AFEQT questionnaires are administered at screening / baseline and at scheduled follow-up (FU) visits. The EQ-5D-5L questionnaire includes 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) assessed with descriptive questions, and a general health score assessed on a Visual Analogue Scale (VAS). For the EQ-5D-5L an index will be derived by comparing the responses to a value set. The index and the health score will each be summarized with mean and standard deviation for randomized arms by visit. The AFEQT questionnaire is a 20-item questionnaire that supports a 4-item symptoms score, an 8-item daily activity score, a 6-item treatment concerns score, and a 2-item treatment satisfaction scale. These are combined into a single AFEQT score. The sub-scores and summary score will be summarized by subject visit and post-procedure assessments, as well as compared between randomized arms using a mixed regression model.
Evaluate post-procedural interventions for atrial arrhythmias | 12 Month and 36 Month
  Post-procedural interventions for atrial arrhythmias will be collected and reported.
Evaluate incidence rate of post-procedure events | 12 Month and 36 Month
  Serious, device-related, and procedure-related adverse events, all-cause and cardio-vascular-related (CV) hospitalizations, all-cause and CV-related mortality, transient ischemic attack and stroke, phrenic nerve palsy, AF-related symptoms and prescription of antiarrhythmic medication will be reported separately.
Characterize AF burden seen on Reveal LINQ | 12 Month and 36 Month
  For subjects in the pilot phase, AF burden will be determined before and after the index ablation from the Cardiac Compass of the Reveal LINQ device.
Characterize AF burden data seen on Reveal LINQ in subjects with any post-procedural intervention for AF | 12 Month and 36 Month
  For subjects in the pilot phase, post-ablation AF burden from the Cardiac Compass of the Reveal LINQ device will be characterized who had a post-procedural intervention for AF.
Comparison of the lesion area as measured by cardiac MRI at Month 3 | 3 Month
  For subjects in the pilot phase, the MRI Core Lab will determine the area of the atrial lesion created by the PVI procedure. Lesion area will be compared between arms of the trial.
Evaluate the relation between outcome and AF burden in the 4 weeks before ablation (Reveal LINQ will be assessed) | 3 Month
  For subjects in the pilot phase, the relation between freedom from AF as assessed for the first primary objective, and the average AF burden from the 4 weeks before the ablation procedure as measured by the Reveal LINQ will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Karl-Heinz Kuck, Prof. Dr., Principal Investigator — Asklepios St. Georg, Hamburg
Locations (5):
- Clinique Pasteur Toulouse, Toulouse, Cedex 3, France
- Germany (4):
  - Herz-Zentrum Bad Krozingen, Bad Krozingen
  - Cardioangiologisches Centrum Bethanien CCB, Frankfurt am Main
  - Asklepios St. Georg, Hamburg
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck, Lübeck